CLINICAL TRIAL: NCT06822192
Title: The Efficacy and Safety of Temporally Interfering in Patients with Disorders of Consciousness
Brief Title: The Temporally Interfering in Patients with Disorders of Consciousness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Doctor, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TI-DOC
Record Dates: First submitted 2025-01-16; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Disorders of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TI (Experimental)
  Interventions: Device: temporally interfering electrical stimulation

INTERVENTIONS:
Device: temporally interfering electrical stimulation — temporally interfering electrical stimulation

SUMMARY:
This project will help the patient recover consciousness by giving TI (temporally interfering) treatment

ELIGIBILITY:
Inclusion Criteria:

In accordance with the international diagnostic criteria for MCS formulated by Giacino in 2002 or the diagnostic criteria for UWS proposed by Laureys in 2010; Patients with disease duration ≥28 days and unconscious improvement tendency in the past one month; No use of any sedative drugs or antiepileptic drugs (sodium or calcium channel blockers) in the past 1 month; stable vital signs; No obvious brain edema, hydrocephalus, and severe brain atrophy; Age from 18 to 70 years old; Informed consent was obtained from the patients' family members.

Exclusion Criteria:

Previous history of neurological or psychiatric disorders; Previous history of traumatic brain injury; History of cancer; Taking sedative drugs or antiepileptic drugs in the past 1 month; Unstable vital signs; Skull defect; The patients' family members did not sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CRS-R (Coma Recovery Scale-revised) | One day before the real/sham stimulus, on the day of the first real/sham stimulus, on the day of the completion of the 10 real/sham stimuli, and 14 days after the completion of the real/sham stimulus
  The CRS-R scale, with scores ranging from 0 to 23, can help to distinguish unresponsive arousal syndrome from micro-conscious states.
Adverse reactions | One day before the real/sham stimulus, on the day of the first real/sham stimulus, on the day of the completion of the 10 real/sham stimuli, and 14 days after the completion of the real/sham stimulus
  Any adverse events related to the study

SECONDARY OUTCOMES:
EEG | One day before the real/sham stimulus, on the day of the first real/sham stimulus, on the day of the completion of the 10 real/sham stimuli, and 14 days after the completion of the real/sham stimulus
  phase-locked values, α, β and other EEG power
fNIRS（functional near-infrared spectroscopy） | One day before the real/sham stimulus, on the day of the first real/sham stimulus, on the day of the completion of the 10 real/sham stimuli, and 14 days after the completion of the real/sham stimulus
  functional connectivity
GOS-E（Glasgow Outcome Scale - Extended） | 2 weeks, 1 month, and 3 months after the end of stimulation
  The outcome of patients was divided into 8 grades by GOS-E, and the higher the grade, the better the prognosis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu Z, Yin L. A mini-review: recent advancements in temporal interference stimulation in modulating brain function and behavior. Front Hum Neurosci. 2023 Sep 14;17:1266753. doi: 10.3389/fnhum.2023.1266753. eCollection 2023. PMID 37780965
- [Background] Yang C, Xu Y, Feng X, Wang B, Du Y, Wang K, Lu J, Huang L, Qian Z, Wang Z, Chen N, Zhou J, Zhang C, Liu Y. Transcranial Temporal Interference Stimulation of the Right Globus Pallidus in Parkinson's Disease. Mov Disord. 2025 Jun;40(6):1061-1069. doi: 10.1002/mds.29967. Epub 2024 Aug 12. PMID 39133053